CLINICAL TRIAL: NCT06026982
Title: Gut Health and the Effect on Substance and Alcohol Cravings
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: City Rescue Mission Medical Clinic (Other)
Responsible Party: Principal Investigator, Anna McCarthy, Principal Investigator, City Rescue Mission Medical Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #23-MCCA-101
Record Dates: First submitted 2023-07-25; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Craving
Keywords: gut health; substance craving; alcohol craving
MeSH Terms: interventions — Probiotics; AT2G25170 protein, Arabidopsis

STUDY DESIGN:
Intervention Model Description: Consent and a pre survey on cravings will be collected. Then participants will take a probiotic/prebiotic and a pickle for 30 days. After 30 days the same survey will be taken by the participants and a paired t test will be used to analyze if there is a statistical change in cravings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gut Health Surveys (Experimental): Participants will take a pre-survey to evaluate their cravings. They will then be started on a regimen of probiotic and prebiotic with a pickle daily for 30 days to improve gut health. Then participants will take the same survey to evaluate if there has been any decrease in cravings.
  Interventions: Dietary Supplement: probiotic and pickle

INTERVENTIONS:
Dietary Supplement: probiotic and pickle — probiotic formula by Rugby Health that has Bacillus Coagulans spores 1billion CFU and inulin 250mg along with a pickle

SUMMARY:
Gut health has been linked with improvement in mental health but no research has been done to evaluate if improving gut health can have an effect on alcohol and substance cravings. This pilot study is to evaluate if any decrease in cravings can be found with probiotics/prebiotics by improving gut health. Participants will take a pre-survey to evaluate their cravings. Participants will then be started on a regimen of probiotic and prebiotic with a pickle daily for 30 days to improve gut health. Then participants will take the same survey to evaluate if there has been any decrease in cravings.

DETAILED DESCRIPTION:
Consent and a pre survey on cravings will be collected. Then participants will take a probiotic/prebiotic and a pickle for 30 days. Participants will be given a probiotic formula by Rugby Health that has Bacillus Coagulans spores 1billion colony forming unit and inulin 250mg along with a pickle daily for 30 days. After 30 days the same survey will be taken by the participants and a paired t test will be used to analyze if there is a statistical change in cravings. Participants will be in a recovery program with a prior history of substance or alcohol abuse and will be abstaining from drugs and alcohol.

The purpose of the study is to evaluate if improving gut health by the above intervention can also decrease substance and alcohol cravings. Probiotics and prebiotics have been shown to improve mental health with a decrease in depression and PTSD but no studies have investigated if improving gut health can decrease substance or alcohol cravings. Probiotics are a cheap intervention that many recovery centers with limited recourses would be able to use. Fermented foods like pickles have been shown to have significant benefit to gut health with improvement in the gut biome. Pickles are also affordable which is why this combination was chosen to be studied.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18-75 years old
* current cravings for substance or alcohol use
* enrolled in a recovery clinic
* able to understand and comply with the requirements of the study
* provision of written informed consent.

Exclusion Criteria:

* Any alcohol or substance use in the past week
* any narcotic use (including methadone and buprenorphine)
* daily probiotic product use in the last 2 weeks
* women who are pregnant or planning to become pregnant during the trial
* if they already have no alcohol or substance cravings
* non English speakers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Decrease in substance or alcohol cravings | 30 days
  Evaluation via the same survey before and after probiotic and a pickle for 30 days to see if there is any change in cravings.
  A pre and post survey will be administered with cravings rated with a scale of 1-5, no cravings would be the number one to extreme cravings with a number of 5. A paired t-test will then be used to analyze the data.

CONTACTS AND LOCATIONS:
Overall Officials: Anna McCarthy, MD MPH, Principal Investigator — City Rescue Mission Medical Clinic

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT06026982/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT06026982/ICF_001.pdf